CLINICAL TRIAL: NCT03896230
Title: Comparison of Ketamine 0.1 mg/kg, 0.2 mg/kg, and 0.3 mg/kg Intravenous Doses for Acute Pain in the Emergency Department: A Prospective, Randomized, Double-blind, Active-controlled, Clinical Trial
Brief Title: Ketamine for Pain in the Emergency Department
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to resource limitations the study was on hold and was then terminated.
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2018-0970
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Acute Pain
Keywords: moderate to severe pain; emergency department patient; ketamine
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: 3 arms each arm getting a different dose of ketamine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study (only the pharmacist supervisor that has no other involvement with the study will know the dose)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: 0.1 mg/kg ketamine (Active Comparator): 0.1 mg/kg in a 100 mL solution of dextrose 5% or sodium chloride 0.9% will be give after patient consent and enrollment in the study, vitals are followed (heart rate, systolic blood pressure and respiratory rate) for 2 hours following completion of ketamine infusion. Evaluated for side effects for 2 hours following completion of ketamine infusion.
  Interventions: Drug: Ketamine Injectable Product
- Arm 1: 0.2 mg/kg ketamine (Active Comparator): 0.2 mg/kg in a 100 mL solution of dextrose 5% or sodium chloride 0.9% will be give after patient consent and enrollment in the study, vitals are followed (heart rate, systolic blood pressure and respiratory rate) for 2 hours following completion of ketamine infusion. Evaluated for side effects for 2 hours following completion of ketamine infusion.
  Interventions: Drug: Ketamine Injectable Product
- Arm 1: 0.3 mg/kg ketamine (Active Comparator): 0.3 mg/kg in a 100 mL solution of dextrose 5% or sodium chloride 0.9% will be give after patient consent and enrollment in the study, vitals are followed (heart rate, systolic blood pressure and respiratory rate) for 2 hours following completion of ketamine infusion. Evaluated for side effects for 2 hours following completion of ketamine infusion.
  Interventions: Drug: Ketamine Injectable Product

INTERVENTIONS:
Drug: Ketamine Injectable Product — Three different doses of ketamine will be administered.

SUMMARY:
This study will prospectively compare the mean Numerical Rating Scale (NRS) pain score reduction amongst three recommended dosing strategies of intravenous ketamine (0.1 mg/kg, 0.2 mg/kg, and 0.3mg/kg) for acute pain in the emergency department (ED).This study will also examine the frequency of adverse events secondary to ketamine including fatigue, dizziness, nausea, headache, feeling of unreality, changes in hearing or vision, mood changes, generalized discomfort, and hallucinations, changes in vital signs. Subgroups for exploratory analysis based on the need for rescue analgesia within two hours of ketamine administration, adequate pain relief, previous opioid tolerance, and age (adults < 65 years old and > 65 years old).

DETAILED DESCRIPTION:
A literature review was performed that searched for randomized clinical trials involving ketamine IV boluses for acute pain in the Emergency Department. Studies involving continuous infusions or intranasal routes of ketamine administration were not included. Thirteen randomized clinical trials were identified meeting this criteria. None of these trials directly compared ketamine doses within the 0.1-0.3 mg/kg range for pain score reduction and adverse events. Many of these trials concluded with the recommendation that further studies were needed to evaluate the optimal dosing of ketamine for acute pain and determine which populations are most ideal for its use. This study will be the first to evaluate ketamine for acute pain in the emergency department at standard of care doses (0.1 mg/kg, 0.2 mg/kg, and 0.3 mg/kg IV) to determine which dose correlates with the most efficacy and safety.

This study will include the following procedures:

* Patient consent, screening, and enrollment will be performed by the treating resident or attending who will remain blinded
* Patient will be assigned a subject number
* Treating resident or attending will notify the ED pharmacist that a patient has been enrolled in the trial
* ED pharmacist will notify the IV room and place the study drug order
* Either the ED pharmacist or a pharmacy supervisor will randomize the subject based on the predetermined randomization list
* Study drug will be prepared as 0.1 mg/kg, 0.2 mg/kg, or 0.3 mg/kg IV dose in a 100 mL solution of dextrose 5% or sodium chloride 0.9%
* ED pharmacist will promptly deliver the study drug to the ED
* Baseline vital signs will be assessed prior to starting the study drug infusion
* Study drug will be administered via IV infusion over 20 minutes
* Treating resident or attending will reassess the patient at 15 minutes from the end of infusion, at 30 minutes from the end of infusion, and then every 30 minutes for up to 120 minutes or until discharge, whichever is sooner

ELIGIBILITY:
Inclusion Criteria:

* Acute pain (including acute on chronic pain)
* Pain score of moderate to severe (> 4/10) on the Numerical Rating Scale
* Provider determines the patient requires intravenous ketamine for analgesia

Exclusion Criteria:

* History of hypersensitivity to ketamine
* Altered mental status
* Psychiatric illness
* Known history of renal or hepatic insufficiency
* Acute head or eye injury
* Suspected intracranial hypertension or mass
* Headache as the chief complaint
* Alcohol or drug abuse
* Received an analgesic within the last four hours
* History of congestive heart failure
* History of aortic or brain aneurysm
* Active Chest Pain
* Porphyria
* Active methadone treatment
* Pregnant or breastfeeding
* Signs of respiratory, hemodynamic, or neurologic compromise

  * Systolic blood pressure < 90 mmHg or > 180 mmHg
  * Heart rate < 50 beats per minute or > 150 beats per minute
  * Respiratory rate < 10 breaths per minute or > 30 breaths per minute
  * Glasgow Coma Score < 15
* Previously received ketamine < 0.3 mg/kg IV for acute pain in the emergency department

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
All study related materials will be kept confidential as required by law. Written documentation and computer files will remain in a locked or password protected location, with access given to those directly responsible for the conduct of the study. In addition, all information will be recorded in such a manner that subjects whose data is included in the analysis cannot be identified directly or through identifiers linked to the subjects.

REFERENCES:
- [Background] Todd KH, Ducharme J, Choiniere M, Crandall CS, Fosnocht DE, Homel P, Tanabe P; PEMI Study Group. Pain in the emergency department: results of the pain and emergency medicine initiative (PEMI) multicenter study. J Pain. 2007 Jun;8(6):460-6. doi: 10.1016/j.jpain.2006.12.005. Epub 2007 Feb 15. PMID 17306626
- [Background] 2. American College of Emergency Physicians Policy Statement. Optimizing the treatment of acute pain in the emergency department. Ann Emerg Med. 2017;70:446-8.
- [Background] Pourmand A, Mazer-Amirshahi M, Royall C, Alhawas R, Shesser R. Low dose ketamine use in the emergency department, a new direction in pain management. Am J Emerg Med. 2017 Jun;35(6):918-921. doi: 10.1016/j.ajem.2017.03.005. Epub 2017 Mar 2. PMID 28285863
- [Background] Crane EH. Highlights of the 2011 Drug Abuse Warning Network (DAWN) Findings on Drug-Related Emergency Department Visits. 2013 Feb 22. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK384680/ PMID 27631059
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] Andolfatto G, Willman E, Joo D, Miller P, Wong WB, Koehn M, Dobson R, Angus E, Moadebi S. Intranasal ketamine for analgesia in the emergency department: a prospective observational series. Acad Emerg Med. 2013 Oct;20(10):1050-4. doi: 10.1111/acem.12229. PMID 24127709
- [Background] Gorlin AW, Rosenfeld DM, Ramakrishna H. Intravenous sub-anesthetic ketamine for perioperative analgesia. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):160-7. doi: 10.4103/0970-9185.182085. PMID 27275042
- [Background] Scheppke KA, Braghiroli J, Shalaby M, Chait R. Prehospital use of i.m. ketamine for sedation of violent and agitated patients. West J Emerg Med. 2014 Nov;15(7):736-41. doi: 10.5811/westjem.2014.9.23229. Epub 2014 Nov 11. PMID 25493111
- [Background] Motov S, Mann S, Drapkin J, Butt M, Likourezos A, Yetter E, Brady J, Rothberger N, Gohel A, Flom P, Mai M, Fromm C, Marshall J. Intravenous subdissociative-dose ketamine versus morphine for acute geriatric pain in the Emergency Department: A randomized controlled trial. Am J Emerg Med. 2019 Feb;37(2):220-227. doi: 10.1016/j.ajem.2018.05.030. Epub 2018 May 16. PMID 29807629
- [Background] Beaudoin FL, Lin C, Guan W, Merchant RC. Low-dose ketamine improves pain relief in patients receiving intravenous opioids for acute pain in the emergency department: results of a randomized, double-blind, clinical trial. Acad Emerg Med. 2014 Nov;21(11):1193-202. doi: 10.1111/acem.12510. PMID 25377395
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884
- [Background] 12. American College of Emergency Physicians. "Sub-Dissociative Ketamine for Analgesia". Policy Resource and Education Paper. November 2017.
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Abbasi S, Bidi N, Mahshidfar B, Hafezimoghadam P, Rezai M, Mofidi M, Farsi D. Can low-dose of ketamine reduce the need for morphine in renal colic? A double-blind randomized clinical trial. Am J Emerg Med. 2018 Mar;36(3):376-379. doi: 10.1016/j.ajem.2017.08.026. Epub 2017 Aug 14. PMID 28821365
- [Background] Bowers KJ, McAllister KB, Ray M, Heitz C. Ketamine as an Adjunct to Opioids for Acute Pain in the Emergency Department: A Randomized Controlled Trial. Acad Emerg Med. 2017 Jun;24(6):676-685. doi: 10.1111/acem.13172. Epub 2017 Mar 22. PMID 28177167
- [Background] Clattenburg EJ, Hailozian C, Haro D, Yoo T, Flores S, Louie D, Herring AA. Slow Infusion of Low-dose Ketamine Reduces Bothersome Side Effects Compared to Intravenous Push: A Double-blind, Double-dummy, Randomized Controlled Trial. Acad Emerg Med. 2018 Sep;25(9):1048-1052. doi: 10.1111/acem.13428. Epub 2018 May 25. PMID 29645317
- [Background] Galinski M, Dolveck F, Combes X, Limoges V, Smail N, Pommier V, Templier F, Catineau J, Lapostolle F, Adnet F. Management of severe acute pain in emergency settings: ketamine reduces morphine consumption. Am J Emerg Med. 2007 May;25(4):385-90. doi: 10.1016/j.ajem.2006.11.016. PMID 17499654
- [Background] Jahanian F, Hosseininejad SM, Amini Ahidashti H, Bozorgi F, Goli Khatir I, Montazar SH, Azarfar V. Efficacy and Safety of Morphine and Low Dose Ketamine for Pain Control of Patients with Long Bone Fractures: A Randomized, Double-Blind, Clinical Trial. Bull Emerg Trauma. 2018 Jan;6(1):31-36. doi: 10.29252/beat-060105. PMID 29379807
- [Background] Mahshidfar B, Mofidi M, Fattahi M, Farsi D, Hafezi Moghadam P, Abbasi S, Rezai M. Acute Pain Management in Emergency Department, Low Dose Ketamine Versus Morphine, A Randomized Clinical Trial. Anesth Pain Med. 2017 Dec 26;7(6):e60561. doi: 10.5812/aapm.60561. eCollection 2017 Dec. PMID 29696126
- [Background] Majidinejad S, Esmailian M, Emadi M. Comparison of Intravenous Ketamine with Morphine in Pain Relief of Long Bones Fractures: a Double Blind Randomized Clinical Trial. Emerg (Tehran). 2014 Spring;2(2):77-80. PMID 26495351
- [Background] Miller JP, Schauer SG, Ganem VJ, Bebarta VS. Low-dose ketamine vs morphine for acute pain in the ED: a randomized controlled trial. Am J Emerg Med. 2015 Mar;33(3):402-8. doi: 10.1016/j.ajem.2014.12.058. Epub 2015 Jan 7. PMID 25624076
- [Background] Motov S, Mai M, Pushkar I, Likourezos A, Drapkin J, Yasavolian M, Brady J, Homel P, Fromm C. A prospective randomized, double-dummy trial comparing IV push low dose ketamine to short infusion of low dose ketamine for treatment of pain in the ED. Am J Emerg Med. 2017 Aug;35(8):1095-1100. doi: 10.1016/j.ajem.2017.03.004. Epub 2017 Mar 3. PMID 28283340
- [Background] Sin B, Tatunchak T, Paryavi M, Olivo M, Mian U, Ruiz J, Shah B, de Souza S. The Use of Ketamine for Acute Treatment of Pain: A Randomized, Double-Blind, Placebo-Controlled Trial. J Emerg Med. 2017 May;52(5):601-608. doi: 10.1016/j.jemermed.2016.12.039. Epub 2017 Mar 6. PMID 28279542
- [Background] 24. Ketalar [package insert]. Chestnut Ridge, NY. Par Pharmaceutical.
- [Background] 25. Food and Drug Administration (FDA). Extended-release (ER) and long-acting (LA) opioid analgesics Risk Evaluation and Mitigation Strategy (REMS). www.fda.gov/downloads/drugs/drugsafety/postmarketdrugsafetyinformationforpatientsandproviders/ucm311290.pdf. Accessed September 20th, 2018.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: 0.1 mg/kg Ketamine | Arm 1: 0.2 mg/kg Ketamine | Arm 1: 0.3 mg/kg Ketamine
Started | 5 | 4 | 2
Completed | 5 | 4 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients that received different doses of ketamine for pain management
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: 0.1 mg/kg Ketamine | Arm 1: 0.2 mg/kg Ketamine | Arm 1: 0.3 mg/kg Ketamine | Total
Number analyzed (Participants) | 5 | 4 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 1 | 9
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 47.4 [28 to 66] | 50.5 [35 to 64] | 68 [64 to 72] | 52.3 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 3 | 1 | 0 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain score using Numerical Rating Scale (NRS) post ketamine infusion. The Numerical Rating Scale (NRS) ranges from 0-to-10 with 0 being no pain and lower numbers representing less pain, so in this case lower numbers will represent better outcomes.
  Pain scores were reported at baseline and then at 15 min/30 min/60 min/90 min and 120 minutes post-infusion.
Time Frame: Within 2 hours post infusion completion
Population: A different number of patients was available for the pain score measurement at the different timepoints. Two patients did not complete infusion, one in the "0.1 mg/kg ketamine" group and one in the "0.3 mg/kg ketamine" group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1: 0.1 mg/kg Ketamine | Arm 1: 0.2 mg/kg Ketamine | Arm 1: 0.3 mg/kg Ketamine
Number analyzed (Participants) | 5 | 4 | 2
score on a scale
  Baseline pain score | 9.4 [9 to 10] | 8.5 [7 to 10] | 7.5 [5 to 10]
  Pain score at 15 min: number analyzed (Participants) | 4 | 2 | 1
  Pain score at 15 min | 5.25 [2 to 9] | 6 [5 to 7] | 2 [2 to 2]
  Pain score at 30 min: number analyzed (Participants) | 4 | 3 | 1
  Pain score at 30 min | 5.25 [2 to 10] | 5.75 [0 to 9] | 6 [6 to 6]
  Pain score at 60 min: number analyzed (Participants) | 4 | 3 | 1
  Pain score at 60 min | 5.25 [2 to 10] | 7 [5 to 9] | 5 [5 to 5]
  Pain score at 90 min: number analyzed (Participants) | 2 | 1 | 1
  Pain score at 90 min | 4.5 [2 to 7] | 7 [7 to 7] | 2 [2 to 2]
  Pain score at 120 min: number analyzed (Participants) | 2 | 0 | 0
  Pain score at 120 min | 4 [3 to 5] |  |

2. Secondary Outcome: Adverse Events
Description: Frequency of adverse events secondary to ketamine including fatigue, dizziness, nausea, headache, feeling of unreality, changes in hearing or vision, mood changes, generalized discomfort, and hallucinations, changes in vital signs.
  Adverse events were reported at baseline and then at 15 min/30 min/60 min/90 min and 120 minutes post-infusion.
Time Frame: Within 2 hours post infusion completion
Population: Number of patients reporting adverse events in the two hours post infusion. Two patients did not complete infusion, one in the "0.1 mg/kg ketamine" group and one in the "0.3 mg/kg ketamine" group and they are not included in the AE reporting.
Measure: Number; unit: participants
Arm/Group | Arm 1: 0.1 mg/kg Ketamine | Arm 1: 0.2 mg/kg Ketamine | Arm 1: 0.3 mg/kg Ketamine
Number analyzed (Participants) | 5 | 4 | 2
participants
  at 15 min post infusion | 2 | 3 | 2
  at 30 min post infusion: number analyzed (Participants) | 4 | 4 | 1
  at 30 min post infusion | 1 | 2 | 1
  at 60 min post infusion: number analyzed (Participants) | 4 | 4 | 1
  at 60 min post infusion | 1 | 2 | 0
  at 90 min post infusion: number analyzed (Participants) | 4 | 4 | 1
  at 90 min post infusion | 1 | 2 | 0
  at 120 min post infusion: number analyzed (Participants) | 4 | 4 | 1
  at 120 min post infusion | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2 hours post infusion.
Description: All adverse events were reported in a systematic manner. A 0-4 scale was used with 0 being "no adverse event" and 4 being "very bothersome adverse event".
Arm/Group | Arm 1: 0.1 mg/kg Ketamine | Arm 1: 0.2 mg/kg Ketamine | Arm 1: 0.3 mg/kg Ketamine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/5 | 3/4 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: 0.1 mg/kg Ketamine (N=5) | Arm 1: 0.2 mg/kg Ketamine (N=4) | Arm 1: 0.3 mg/kg Ketamine (N=2)
Dizziness (General disorders) | 2 (3) | 3 (5) | 1 (2) — A scale 0-4 was used to describe dizziness with 0 being "no dizziness" and 4 being "very bothersome" dizziness.
Changes in vision (Eye disorders) | 1 (5) | 1 (1) | 1 (1) — A scale 0-4 was used to changes in vision with 0 being "no changes" and 4 being "very bothersome" changes.
Generalized discomfort (General disorders) | 2 (5) | 2 (7) | 2 (3) — A scale 0-4 was used to generalized discomfort with 0 being "no generalized discomfort" and 4 being "very bothersome" generalized discomfort.
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — A scale 0-4 was used to measure headache with 0 being "no headache" and 4 being "very bothersome" headache.
Unreality (General disorders) | 1 (1) | 3 (7) | 2 (3) — A scale 0-4 was used to measure unreality with 0 being "no unreality" and 4 being "very bothersome" unreality.
Fatigue (General disorders) | 1 (3) | 2 (6) | 0 (0) — A scale 0-4 was used to measure fatigue with 0 being "no fatigue" and 4 being "very bothersome" fatigue.
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) — A scale 0-4 was used to measure nausea with 0 being "no nausea" and 4 being "very bothersome" nausea.
Mood change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — A scale 0-4 was used to measure mood change with 0 being "no mood change" and 4 being "very bothersome" mood change.
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2) — A scale 0-4 was used to measure hallucination with 0 being "no mood Hallucination" and 4 being "very bothersome" hallucination.

LIMITATIONS AND CAVEATS:
The study was initiated in 2019 and was then put on hold because of COVID. Post-COVID, the study was opened to enrollment again but due to limited resources and lack of enrollment, the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03896230/Prot_SAP_001.pdf